CLINICAL TRIAL: NCT03070587
Title: Effect of Mindfulness and Loving Kindness Meditation on Symptoms of Social Anxiety Disorder
Brief Title: A Pilot Study of Loving-Kindness Meditation for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Komazawa University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Social Anxiety Disorder; Compassion
MeSH Terms: conditions — Phobia, Social | interventions — Sagittal Abdominal Diameter

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Affect Training for SAD (Experimental): The intervention will be conducted in groups with 68 participants and 2 facilitators/therapists per group. The groups will meet once a week for 12 successive weeks and each session will be approximately 60 minutes long.
  Interventions: Behavioral: Positive Affect Training for SAD
- Wait list Control (No Intervention): These participants will not be given an intervention until after they have completed the study.

INTERVENTIONS:
Behavioral: Positive Affect Training for SAD — The PAT-S protocol will teach the participants the basics of mindfulness and how to be aware of their physical sensation, thoughts, and emotion at present moment by a nonjudgmental way in breathing, standing, or eating. After two mindfulness sessions, lovingkindness meditation (LKM) will be introduced. The participants will be taught to identify and focus the positive feelings such as gratitude, love, kindness, peacefulness, or friendliness when they wish their benefactor and beloved ones who they feel grateful or respectful, and transfer these feelings first to themselves, then to a neutral individual, to people whom they dislike, and finally to all living beings.
  Arms: Positive Affect Training for SAD

SUMMARY:
The purpose of this study is to develop and test a mindfulness and loving-kindness based intervention, Positive Affect Training (PAT), to enhance positive affect such as compassion, love, and gratitude and reduce symptoms of social anxiety disorder (SAD). PAT involves a combination of practicing mindfulness meditation and loving kindness meditation in groups. Although PAT has been shown to be effective for dysthymic disorder, one area that remains unclear is whether the PAT protocol for SAD can address the social anxiety symptoms in Japanese adults with SAD. The goal of the research is to test the initial feasibility and efficacy in increasing positive affect and decreasing negative affect in individuals recruited from the general community who are social anxious. If PAT is also effective for Japanese SAD patients, it could be more cost-effective and noninvasive option to address social anxiety disorder.

DETAILED DESCRIPTION:
Mindfulness based stress reduction (MBSR) and mindfulness based cognitive therapy (MBCT), which are based on Buddhist tradition, has been shown to be effective for many psychological disorders including anxiety disorders. Buddhist tradition, however, has many kinds of meditation which would be able to address psychological distress but MBSR and MBCT has not focused. Loving kindness meditation (LKM) is one of promising meditation to be effective for psychological disorders because it is designed to increase feelings of social connection and compassion for one's self and others, whose focus is different from mindfulness meditation. Since mindfulness meditation is designed to observe and accept current internal experiences as they are while maintaining a primary focus on the breath sensations, it would cultivate less compassion than LKM would. Because patients with SAD tend to be self-critical, cultivating compassion for self and others with LKM would be more effective to reduce symptoms of SAD than MBSR and MBCT. In support of the view that KM increases positive mood and a sense of connection and positivity towards others, previous studies with non-clinical samples, schizophrenia, dysthymia, and PTSD had decreased the mental illness. The intervention protocol that the investigators plan to use was developed by Dr. Kearney and Dr. Hofmann. The PAT protocol has been shown to generate positive, and attenuating negative affect in patients with PTSD and mood disorder. The investigators aim to test the initial efficacy of PAT in individuals with SAD. The investigators hypothesize the intervention would show significant improvement in subjects' self-reported ratings of negative and positive affect and the brain asymmetry. Dr. Hofmann, a prominent researcher and clinical psychologist who is the foremost expert in LKM will serve as a collaborator. Dr. Kaiya, a Japanese CBT therapist for anxiety disorders will serve as an outside consultant for the study.

ELIGIBILITY:
Inclusion Criteria:

Must be at least 20 years of age Responds positively to the question on the recruitment material (flyer and posting): "Have you been feeling anxious or distressed in social situations?" Must be diagnosed with Social Anxiety Disorders using the DSM-5 criteria Must have SAD as the primary diagnosis according to DSM-5 criteria Must have a negative affect scale score of the LSAS of at least 30 (a cutoff point which SAD is unlikely)

Exclusion Criteria:

Participants who are at risk of harming themselves will be excluded from participating in the study. Suicidality will be assessed after obtaining consent during the screening visit. In addition, the Beck Depression Inventory will be examined for self-reported suidicality. If a participant is found to have suicidal ideation (i.e., exceed a score of 2 on the suicide item of BDI-II), the principal investigator will be contacted immediately and appropriate follow-up care will be provided by referring the participant to the emergency room.

Participants will be assessed through a screening interview using the Structured Clinical Interview for DSM-5 for disorders that could impose a safety risk for the participants or others (e.g., bipolar disorder, schizophrenia, etc). Subjects who endorse "yes" responses to the screening items will be excluded.

Participants who are receiving any psychiatric or psychological treatment for any psychological disorders at the time of the assessment will be excluded from the study. Participants who initiate such treatments while being enrolled in the study will be closely monitored. These participants will be allowed to remain in the study, but will later be excluded from the data analyses. They are allowed to remain in the study for ethical reasons.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Liebowitz Social Anxiety Scale (LSAS) | Baseline and 6 months
  A self-report measure that assesses symptoms of distress experienced when socializing with others.

SECONDARY OUTCOMES:
Change from Baseline in Self-Compassion Scale (SCS) | Baseline and 6 months
  Participants rated a 26-item test using 5-point scale that ranges from "almost never" (1) to "almost always" (5). Items are averaged, yielding a range from 1 to 5.
Change from Baseline in Positive and Negative Affect Scale (PANAS) | Baseline and 6 months
  Participants in the PANAS are required to respond to a 20-item test using 5-point scale that ranges from very slightly or not at all (1) to extremely (5). The total range is from 1 to 100.
Change from Baseline in compassion subscale of Differential Positive Emotions Scale | Baseline and 6 months
  Participants in the DPES are required to respond to a 38-item test using 7-point scale that ranges from "strongly disagree" (1) to "strongly agree" (7). Items are averaged, yielding a range from 1 to 7.

CONTACTS AND LOCATIONS:
Overall Officials: Kohki Arimitsu, Ph.D., Principal Investigator — Kwansei Gakuin University
Locations (1):
- Kwansei Gakuin University, Nishinomiya, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofmann SG, Petrocchi N, Steinberg J, Lin M, Arimitsu K, Kind S, Mendes A, Stangier U. Loving-Kindness Meditation to Target Affect in Mood Disorders: A Proof-of-Concept Study. Evid Based Complement Alternat Med. 2015;2015:269126. doi: 10.1155/2015/269126. Epub 2015 Jun 1. PMID 26136807
- [Background] Hofmann SG, Grossman P, Hinton DE. Loving-kindness and compassion meditation: potential for psychological interventions. Clin Psychol Rev. 2011 Nov;31(7):1126-32. doi: 10.1016/j.cpr.2011.07.003. Epub 2011 Jul 26. PMID 21840289
- [Background] Arimitsu K, Hofmann SG. Effects of compassionate thinking on negative emotions. Cogn Emot. 2017 Jan;31(1):160-167. doi: 10.1080/02699931.2015.1078292. Epub 2015 Sep 11. PMID 26362245
- See also: The detailed information web-site — https://clinical-affective-science.org/LKM.html